CLINICAL TRIAL: NCT04906252
Title: Ventricular Fibrillation and Electrocardiographic Rhythm vs Echocardiographic Rhythm During Cardiac Arrest
Brief Title: Vfib by ECG or Echo During Cardiac Arrest
Acronym: REASON3-2021
Status: Completed | Type: Observational
Sponsor: Romolo Gaspari (Other)
Collaborators: Temple University (Other); Stony Brook University (Other); University of Ottawa (Other); ChristianaCare (Other); Boston Medical Center (Other); Dartmouth College (Other); University of Alabama at Birmingham (Other); University of Rochester (Other); Baystate Medical Center (Other); Medical College of Wisconsin (Other); University of Pennsylvania (Other); Prisma Health-Midlands (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); Staten Island University Hospital (Other); State University of New York - Upstate Medical University (Other); University of Manitoba (Other); Mayo Clinic (Other); Kaweah Delta Health Care District (Other); SBH Health System (Other); Yale University (Other); Johns Hopkins University (Other); The University of Texas at San Antonio (Other); Wake Forest University Health Sciences (Other); University of Arkansas (Other); Valleywise Health (Other); Kendall Healthcare Group, Ltd. (Industry); Truman Medical Center (Other); Oregon Health and Science University (Other); Vassar Brothers Medical Center (Other); Brookdale University Hospital Medical Center (Other); University of Kansas Medical Center (Other); University of Maine (Other); University of Colorado, Denver (Other); Duke University (Other); University at Buffalo (Other); North Shore University Hospital (Other); Hartford Hospital (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Florida (Other); University of Maryland (Other); Sutter Medical Foundation (Other); Arizona School of Health Sciences (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor-Investigator, Romolo Gaspari, Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H00021832
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest
Keywords: Echocardiography; Ultrasound; Ventricular Fibrillation; Vfib
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation | interventions — Echocardiography; Ultrasonography; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ventricular Fibrillation: Patients presenting to the Emergency Department after out of hospital cardiac arrest demonstrating Ventricular Fibrillation (Vfib) Cardiac Arrest or Patients demonstrating Vfib during cardiac arrest.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Electrocardiogram (ECG)
- PEA: Patients presenting to the Emergency Department after out of hospital cardiac arrest demonstrating Pulseless Electrical Activity (PEA) Cardiac Arrest. Patients demonstrating PEA during cardiac arrest
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Electrocardiogram (ECG)
- Asystole Cardiac Arrest: Patients presenting to the Emergency Department after out of hospital cardiac arrest demonstrating Asystolic Cardiac Arrest. Patients demonstrating Asystole during cardiac arrest
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Electrocardiogram (ECG)

INTERVENTIONS:
Diagnostic Test: Echocardiography — Patients presenting in cardiac arrest will undergo echocardiography as is the standard of care at their institution
  Other Names: Ultrasound
Diagnostic Test: Electrocardiogram (ECG) — Patients presenting in cardiac arrest will undergo an electrocardiogram (ECG) as is the standard of care at their institution

SUMMARY:
The goal of this study is to measure survival rates associated with patients presenting in cardiac arrest based on their electrocardiographic rhythm and their echocardiographic rhythm. Electrocardiographic rhythm is defined as the rhythm on the ECG and echocardiographic rhythm is the rhythm visualized on bedside ultrasound. Specifically, we will categorize patients based on identical rhythms and dichotomous rhythms with an interest in outcomes in the patient group where their echocardiographic and electrographic rhythms do not match. This is important as current ACLS protocols use electrocardiographic rhythms to determine therapy but limited research implies that therapeutic decisions based on echocardiographic rhythm may produce increased survival.

This study will occur during emergency department resuscitation of patients presenting in cardiac arrest. Patients presenting to the emergency department after cardiac arrest will undergo standard resuscitation based on ACLS protocols. Ultrasound imaging will be performed as soon as possible after the patient arrives and digitally recorded, as is currently the standard of care at the institute. Simultaneous recording of the ECG rhythm strip will occur as well. This will be repeated for as many pauses in CPR as is warranted.

Each site will record data based on the Utstein nomenclature including patient demographics, arrest details and survival outcomes. Ultrasound images and ECG recordings will be de-identified and submitted to a central database. Data will be uploaded into a centralized database. Statistical analysis will analyze outcomes based on echocardiographic and sonographic findings. Our aim is to measure the survival benefit of treating out of hospital cardiac arrest using echocardiographic rhythm instead of electrocardiographic rhythm.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational trial involving sites across the United States and Canada. Patients will be enrolled through the emergency department either presenting in cardiac arrest, or going into cardiac arrest while in the emergency department after having arrested out of hospital. Advanced Cardiac Life Support (ACLS) protocols and institutional policies for resuscitation will be followed, as is the current standard of care. A patient encounter will conclude upon halting of cardiopulmonary resuscitation. Patient outcome will be evaluated by chart review or follow-up.

Programs involved in this study must have already integrated echocardiography into Cardiac Arrest clinically and have established procedures for how imaging is performed in the context of CPR. Echocardiography will not hinder or impair resuscitative efforts in any way, including halting CPR or prolonging pauses in CPR. Sonographic images will be obtained during designated pauses in chest compressions, as is routine care, during CPR for pulse checks, rhythm checks, and necessary resuscitative procedures.

Echocardiography will be performed as appropriate to obtain diagnostic information for each particular patient during resuscitative efforts. Recording of the image loops will be performed during image acquisition according to standard technology availability and clinical protocols at each site. To facilitate image acquisition, the ultrasound probe may be placed in the epigastrium or parasternal region during CPR with the heart centered in the field of view, if it will not interfere with ongoing resuscitation. Recording of the images can begin immediately upon pauses of CPR using whatever means are available at the site. Sonographic images will be obtained by competent personnel with experience in bedside cardiac ultrasound. This information will be made available to the physician taking care of the patient.

Continuous ECG tracings are displayed during cardiac arrest, and for the purpose of this study recordings of these ECG tracings will need to be digitally recorded. These digital ECG 'rhythm strips" will be matched with contemporaneous recordings of the ultrasound images of the heart.

Subject data, with identifiers removed, will be uploaded into the REDcap web-based database. Data will be obtained from initial patient encounter, patient records, and EMS records when available.

Contemporaneous digital recordings of ultrasound images and ECG rhythm strips blinded to patient identifiers will be included in a centralized database. Echocardiographic images will be reviewed and interpreted by the central coordinating site blinded to patient information. ECG images will be reviewed and interpreted by the central coordinating site blinded to patient information.

Patient cohorts will be compared for the electrical activity by ECG and the myocardial activity by echo.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting in out-of-hospital, atraumatic cardiac arrest

Exclusion Criteria:

* Resuscitation ended due to end of life decisions
* Documented allergy to ultrasound gel
* Technical malfunction of ultrasound machine during imaging that prevents use Ultrasound machine unable to record images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting after out of hospital cardiac arrest to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Survival to Hospital Admission | up to 60 minutes
  Percentage of patients who survive at the point where they are admitted to the hospital
Rhythm Change post defibrillation | up to 60 minutes
  Percentage of patients who when defibrillated have a change in their cardiac rhythm as reflected by Electrocardiogram (ECG) report

SECONDARY OUTCOMES:
Return of Spontaneous Circulation (ROSC) | up to 60 minutes
  Percentage of patients who demonstrate return of spontaneous circulation (ROSC)
Survival to Hospital Discharge | up to discharge, on average 7 days
  Percentage of patients who survive at the point where they are discharged from the hospital
Ventricular Fibrillation (VFib) detected via Ultrasound but not detected via Electrocardiogram (ECG) | up to 60 minutes
  The percentage of patients with Ventricular Fibrillation (VFib)which is detected via ultrasound examination but is not detected via Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, PhD, Principal Investigator — UMass Medical School
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Stony Brook University, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Allegheny Hospital, Pittsburgh, Pennsylvania
  - Univesity of Texas San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
As a cardiac arrest study, there is not a current plan to share individual data but this may be reconsidered if required